CLINICAL TRIAL: NCT00478517
Title: Treatment With Erythropoetin in Patients With Spinal Trauma With Neurological Deficit, Maximum Tolerated Dose Study. TETRAM2
Brief Title: TETRAM 2. Treatment With Erythropoetin in Patients With Spinal Trauma With Neurological Deficit, Maximum Tolerated Dose Study
Acronym: TETRAM2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2006.455
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Spinal Trauma With Neurological Deficit
Keywords: Spinal trauma; erythropoietin; dose escalation study
MeSH Terms: interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Erythropoetin (rHuEPO, EPREX®)

SUMMARY:
The social, psychological, economic burden of Spinal trauma with deficit is great, and there is no curative treatment.

Erythropoetin (EPO) is promising, due to its neuroprotective effects demonstrated in vitro, in vivo in animal models and in a preliminary study including patients with stroke.

The study primary end point is to find out the maximum tolerated dose of EPO. This is based on the occurrence of pulmonary embolism during a 14 day delay following EPO injection. Secondary end points include comparisons of EPO kinetics in blood and cerebrospinal fluid (CSF), study of EPO effects on several inflammatory and apoptotic bio markers and blood cell counts.

The experimental design is a dose scale study (600 to 2400 UI/Kg), using a single dose of rHuEPO, (EPREX®). The EPO dose is defined using a Bayesian continuous reassessment Method (CRM). The sample size is expected for less than 20 patients.

Eligible patients are patients aged 15 to 65 years, able to receive the EPO injection within 12 hours of a spinal trauma, without vital blood loss or associated diseases. The follow-up lasts 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 15 to 65 years, covered by a social insurance system, having given an informed consent (or attested by a third person if unable to sign, or parents consent in minors), within 12 hours of a spinal trauma, without vital organ deficiency from a non spinal origin

Exclusion Criteria:

* Impaired consciousness,
* Treatment not given within 12 hours,
* Cervical arthritis,
* Respiratory failure requiring artificial ventilation,
* Patient requiring blood transfusion superior to 2 units,
* Uncontrolled severe hypertension,
* Unstable hemodynamics,
* Patient suffering from epilepsy,
* Recent or uncontrolled angina pectoris,
* Having received high doses of glucorticoïds,
* Pregnant or breasting,
* With more than 15 g/ml of haemoglobin,
* With previous thrombo embolism disease,
* With allergy to Low molecular Weight heparin, or
* Participating in another interventional study

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2007-05

PRIMARY OUTCOMES:
Pulmonary embolism occurring during a 14 day delay following EPO injection.

SECONDARY OUTCOMES:
Blood cells count biomarkers of inflammation and apoptosis: measured at Day 0 (Epo antibodies) D1, D3 and D 14 ICAM-1 Fas-Ligant M-30 IL-10 in blood and CSF. Clinical ASIA score, morbi-mortality Evolution of spinal MRI between D0 and D28.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lieutaud, MD, Principal Investigator — Hospices Civils de Lyon